CLINICAL TRIAL: NCT04036513
Title: Split Mouth Comparison of Minimally Invasive Non Surgical Therapy Versus Conventional Scaling and Root Planing for Treatment of Periodontitis
Brief Title: Minimally Invasive Non Surgical Therapy Versus Conventional Scaling and Root Planing for Treatment of Periodontitis
Acronym: MINST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ljubljana (Other)
Responsible Party: Principal Investigator, Rok Gašperšič, Assist. Prof., University of Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-1-1
Record Dates: First submitted 2019-07-25; First posted 2019-07-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Periodontal Diseases
Keywords: Periodontitis; MINST; Scaling and root planing; Split mouth; 3D analysis
MeSH Terms: conditions — Periodontal Diseases; Periodontitis

STUDY DESIGN:
Intervention Model Description: Split mouth - experimental and control side in the same individual Side selection will be randomized
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Evaluator different to care provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MINST (Experimental): Usage of magnification loupes, specific thin and delicate tips together with piezoelectric device and specifically designed Hu-Friedy "mini five", "micro mini five", and "after five" Gracey curettes under local anaesthesia.
  Interventions: Procedure: MINST
- Conventional SRP (Active Comparator): Conventional non-surgical mechanical treatment using piezoelectric device (PiezoLED, Kavo) and standard Gracey curettes under local anaesthesia.
  Interventions: Procedure: Conventional SRP

INTERVENTIONS:
Procedure: MINST — For reducing the need of surgical treatment in patients with chronic periodontal disease, we will use specifically designed Hu-Friedy curettes "mini five", "micro mini five" and "after five" together with piezoelectric device with thin and delicate tips that produce less periodontal trauma than usual Gracey curettes.
  Arms: MINST
Procedure: Conventional SRP — Scaling and root planing with conventional instruments.
  Arms: Conventional SRP

SUMMARY:
Minimally invasive non-surgical therapy (MINST) is a new approach towards regeneration of deep periodontal defects. Important part of MINST procedure, besides usage of magnification loupes and piezo-electric devices seems to be the usage of special mini-curettes, originally mini-five and after mini-five of Hu-Friedy. So far only descriptive data about the clinical effects of such procedure are available and comparative studies that would include other treatment alternatives are lacking. Therefore, the aim of our study is, on split-mouth model, to compare the number of diseased sites (defined by probing depth ˃ 4 mm and bleeding on probing) after conventional non-surgical therapy and MINST with the usage of special mini-curettes. In addition, new 3D parameters obtained from 3D optical scanning will be developed for evaluation of volume changes of soft tissues.

ELIGIBILITY:
Inclusion Criteria:

* periodontitis Stage III, grade B/C
* at least 20 teeth
* at least 9 teeth (excluding molars) in the upper jaw
* without FPD, implants
* without occlusal trauma signs
* no pathology of endodontic origin
* without chronic systemic diseases
* no periodontal treatment in the last 6 months

Exclusion Criteria:

* poor oral hygiene (PI > 20% at evaluation)
* antibiotic treatment in the last 6 months or during the observation period
* pregnant women, lactation, serious chronic systemic diseases, medication with known influence on periodontium or wound healing

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2021-04-02 (Actual); Study Completion 2021-04-02 (Actual)

PRIMARY OUTCOMES:
Number of diseased sites | 3 months, 6 months, 12 months
  Difference in No of Sites with PPD (probing pocket depth) > 4 mm and BOP (bleeding upon probing)

SECONDARY OUTCOMES:
PPD | 3 months, 6 months, 12 months
  Average probing pocket depth
CAL | 3 months, 6 months, 12 months
  Clinical attachment loss
REC | 3 months, 6 months, 12 months
  Gingival recession
VOL | 1 week, 1 month, 3 months, 6 months, 12 months
  Volumetric 3D differences evaluated by optical scanning

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No
Have no intention to share

REFERENCES:
- [Background] Nibali L, Yeh YC, Pometti D, Tu YK. Long-term stability of intrabony defects treated with minimally invasive non-surgical therapy. J Clin Periodontol. 2018 Dec;45(12):1458-1464. doi: 10.1111/jcpe.13021. Epub 2018 Nov 5. PMID 30307641
- [Background] Nibali L, Pometti D, Chen TT, Tu YK. Minimally invasive non-surgical approach for the treatment of periodontal intrabony defects: a retrospective analysis. J Clin Periodontol. 2015 Sep;42(9):853-859. doi: 10.1111/jcpe.12443. Epub 2015 Sep 29. PMID 26257238
- [Derived] Kucic AC, Gaspersic R. Minimally invasive non-surgical therapy (MINST) in stage III periodontitis patients: 6-month results of a split-mouth, randomised controlled clinical trial. Clin Oral Investig. 2023 May;27(5):2075-2087. doi: 10.1007/s00784-023-04994-4. Epub 2023 Apr 4. PMID 37014505